CLINICAL TRIAL: NCT03519230
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Multicenter Trial of Maintenance Treatment With BGB-290 Versus Placebo in Patients With Platinum-sensitive Recurrent Ovarian Cancer
Brief Title: Maintenance Treatment With BGB-290 Versus Placebo in Participants With Platinum-sensitive Recurrent Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGB-290-302; ChiCTR1800014643 (Registry Identifier: Chinese Clinical Trial Registry); CTR20171666 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2018-04-26; First posted 2018-05-08 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pamiparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental)
  Interventions: Drug: Pamiparib capsule
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Pamiparib capsule — 60 mg twice daily (BID), orally (per os-PO)
  Other Names: BGB-290
  Arms: Treatment arm
Drug: Placebo capsule — 60mg BID, PO
  Arms: Placebo arm

SUMMARY:
To evaluate the efficacy, safety and tolerability of maintenance therapy with BGB-290(Pamiparib) versus placebo in Chinese participants with recurrent ovarian cancer who achieved a complete response (CR) or partial response (PR) after platinum-based chemotherapy

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically diagnosed high-grade serous or endometrioid ovarian cancer (including primary peritoneal and fallopian tube cancer)
2. Completion of ≥2 previous platinum-containing regimens (eg, carboplatin or cisplatin)
3. Complete response (CR) or partial response (PR) achieved with last platinum-based chemotherapy regimen as determined by investigator per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
4. Ability to be randomized ≤8 weeks after last dose of platinum

Key Exclusion Criteria:

1. Prior treatment with a poly (ADP-ribose) polymerase (PARP) inhibitor
2. Progressive disease (PD) as per CA-125 criteria before randomization
3. Diagnosis of myelodysplastic syndrome (MDS)
4. Known history of intolerance to the excipients of the Pamiparib capsule

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) by blinded Independent Review Committee (BIRC) assessment | up to 8 years

SECONDARY OUTCOMES:
Overall survival | up to 9 years
Objective response rate by investigator assessment | up to 2 years
Duration of response by investigator assessment | up to 2 years
PFS by investigator assessment | up to 8 years
Time to response by investigator assessment | up to 8 years
Number of participants with treatment-emergent adverse events (TEAEs) | up to 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (28):
- China (28):
  - Anhui Provincial Cancer Hospital Aka West Branch of Anhui Province Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Maternal and Child Health Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Second University Hospital, Chengdu, Sichuan
  - Tianjin Central Hospital of Gynecology Obstetrics, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/